CLINICAL TRIAL: NCT06554990
Title: Effect of Sensory-Perceptual Motor Training on Activities of Daily Living and Hand Functions in Unilateral Cerebral Palsy
Brief Title: Sensory Perceptual Training on Activities of Daily Living and Hand Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, hanaa mohsen, Associate professor, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hanaa M
Record Dates: First submitted 2024-08-09; First posted 2024-08-15 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Palsy, Spastic
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Other): physical therapy excersises
  Interventions: Other: physical therapy excersies
- intervention (Experimental): sensory perceptual training
  Interventions: Other: sensory perceptual motor exercises

INTERVENTIONS:
Other: physical therapy excersies — 1- selected physical therapy exercises
  Arms: control
Other: sensory perceptual motor exercises — selected sensory perceptual motor exercises
  Arms: intervention

SUMMARY:
Many risk factors can come to the fore in CP. With the new studies on CP, new risk factors are defined and existing risks are better understood. In the light of current information, general risk factors for CP are defined as premature birth, fetal growth restriction, multiple pregnancies, infections in the fetal or neonatal period, birth asphyxia, perinatal stroke, and congenital developmental disorders In addition, related risk factors are classified as prenatal, perinatal and postnatal

DETAILED DESCRIPTION:
Children and youth with cerebral palsy face unique challenges when learning, practicing, and mastering activities of daily living (ADLs). Active participation in dressing, feeding, toileting, clothing management, and small space mobility is influenced by body structures and function and environmental and personal factors

ELIGIBILITY:
Inclusion Criteria:

* Modified Ashworth 1 and 1 +
* GMFCS level I and II
* Able to understand and follow instructions

Exclusion Criteria:

* fixed contracture or deformities in the spine or extremities
* visual or respiratory Problems,
* orthopedic surgery

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Katz Index | pre and post treatment for 12 weeks
  It was especially designed to evaluate activities of daily living

SECONDARY OUTCOMES:
Jebsen Taylor Hand Function Test | pre and post treatment for 12 weeks
  It was especially designed to evaluate Time motor performance
box and block test | pre and post treatment for 12 weeks
  It was especially designed to evaluate the gross manual dexterity

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa mohsen, Principal Investigator — Associate professor
Locations (2):
- Egypt (2):
  - Badr UNIVERSITY and Cairo University, Cairo
  - BADR, Cairo

IPD SHARING:
Plan to Share IPD: No